CLINICAL TRIAL: NCT01651819
Title: Effects of Physiotherapy in the Treatment of Neurogenic Bladder in Patients Infected With Human T-Lymphotropic Virus 1
Brief Title: Urological Physical Therapy in HTLV-1 With Urinary Symptoms
Acronym: UROHTLV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, ROSANA CRISTINA PEREIRA DE ANDRADE, coordenadora do Ambulatório de Fisioterapia Nas Disfunções perineias, Hospital Universitário Professor Edgard Santos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROAND2012
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Tropical Spastic Paraparesis; HTLV-1
Keywords: HTLV-1; neurogenic bladder; physical therapy; Tropical Spastic Paraparesis
MeSH Terms: conditions — Paraparesis, Tropical Spastic; Urinary Bladder, Neurogenic | interventions — Electric Stimulation Therapy; Behavior Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urological physical therapy (Experimental): Urologic physical therapy is going to be apply in 20 patients with HTLV-1 infection and overactive bladder symptoms like urgency, incontinence and nocturia. There will be 20 sessions with one hour duration and a interval of 3 or 4 days between the sections.
  Interventions: Procedure: Urological physical therapy

INTERVENTIONS:
Procedure: Urological physical therapy — Individual patient attending with one hour duration beginning with Behavior therapy and education, teaching urinary maneuvers, water adequate intake. Second part is manual therapy an Kinesiotherapy with specific exercises, followed by patient repetition. Last part is constituted by electrotherapy for specific muscle stimulation and biofeedback.
  Other Names: Electrotherapy;; Behavior therapy;; Manual therapy;; Kinesiotherapy.

SUMMARY:
Urological physical therapy is described to improve urinary symptoms in patients with myelopathy or neurological dysfunction and to increase the quality of life. Although it was never tested on HTLV-1 associated overactive bladder syndrome, an disabling disease that is common seen in HAM/TSP patients but can also appear as an isolated form. Our hypothesis is that urological physical therapy can improve urinary symptoms like incontinence, urgency and nocturia in HTLV-1 infected population with those complains.

DETAILED DESCRIPTION:
The T-lymphotropic virus type 1 (HTLV-1) is an human retrovirus that was proved to be the main agent of the acute T cell lymphoma/leukemia (ATLL) and a progressive neurological disease called HTLV-1 associated myelopathy/ tropical spastic paraparesis (HAM/TSP).

The HTLV-1 was first isolated in 1980 and it is endemic in Japan, Caribbean, Africa and South America. It is estimated that about 20 million people is infected worldwide. In Brazil it is present in all states with variable prevalences. The factors associated with HTLV-1 transmission in Brazil are related to the social and demographic condition, characterized by rural exodus and increase of urban population in the coast areas.

Several studies based in Brazil reported that the epicenter of HTLV-1 infection is on Bahia, Maranhão and Pernambuco with the highest prevalence of 1,8% in Salvador, Bahia capital.

The urinary incontinence is a bladder-sphincter disturbance often found in HTLV-1 patients. In this infection the most common pathology finding is overactive bladder syndrome due detrusor overactivity and sphincter-detrusor dyssynergia and the symptoms are urgency, nocturia and incontinence.

This disabling disease is associated with psychosocial issues like loss of self confidence, social isolation and reduced quality of life.

The physical therapy treatment have the objective of promote social adequacy and reestablish the bladder function. It is based on resources like: bladder reeducation, biofeedback, kinesiotherapy of the pelvic wall, utilization of vaginal cones and electrostimulation.

Those can be associated or not with anticholinergic drugs and bladder catheterization.

The need of urologic and gynecologic physical therapy follow up in patients with HTLV-1 and neurogenic bladder is important to reduce disability, preserve pelvic muscles and renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HTLV-1 with more than 18 years and neurogenic bladder defined by urodynamic study.

Exclusion Criteria:

* Diabetes Mellitus,
* Stroke,
* Multiple Sclerosis,
* Parkinson disease,
* use of pacemaker,
* urinary infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Reduction in urinary symptoms | 6 months
  reduce or cure the complaints of urinary symptoms measured by daily and nocturnal frequency, presence of incontinence, urgency, dysuria.

SECONDARY OUTCOMES:
Improve in quality of life | 6 months
  improving the quality of life measured by King' Health scale that is applied before and after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rosana Andrade, Master, Principal Investigator — Federal University of Bahia
Locations (1):
- Hospital Universitário Prof. Edgard Santos, Salvador, Estado de Bahia, Brazil